CLINICAL TRIAL: NCT04700020
Title: (Partial) Empty Sella - Incidental Finding or the Cause of Hormonal Dysregulation?
Brief Title: An Assessment of the Occurrence of Hormone Deficiency in Patients With Empty Sella
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019/119
Record Dates: First submitted 2021-01-05; First posted 2021-01-07 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2020-12

CONDITIONS: Empty Sella
MeSH Terms: conditions — Empty Sella Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients above the age of 18 years (Other): In the context of this study, we will take two blood samples. In addition to the second blood sample, an insulin tolerance test (ITT) is also performed, even if the result of the blood values is normal.
  MRI will only be performed if the previous imaging was done more than two years ago or when the quality of the MRI was not good enough to measure the volume of the pituitary gland.
  Interventions: Diagnostic Test: ITT

INTERVENTIONS:
Diagnostic Test: ITT — In the context of this study, we will take two blood samples. In addition to the second blood sample, an insulin tolerance test (ITT) is also performed, even if the result of the blood values is normal. MRI will only be performed if the previous imaging was done more than two years ago or when the quality of the MRI was not good enough to measure the volume of the pituitary gland. This is needed for better analysis of the pituitary gland, as the pituitary volume could be important for the hormonal abnormalities.
  Other Names: MRI; Blood Withdrawal

SUMMARY:
The goal of this prospective study is to analyse the hormonal components in the blood of patients that were diagnosed with empty sella. Hereby we only take the hormones into consideration that are produced by the pituitary gland and/or are influenced by it due to positive/negative feedback. These are GH, ACTH, TSH, FSH, LH, PRL, oxytocine, ADH but also IGF-1, estradiol, testosteron, F4 and cortisol. The purpose is to see if abnormalities of the blook levels can be explained by the absence/shrinking of the pituitary gland. During this study, there will be a blood draw twice. The reason is to avoid wrong positive and negative results. Together with the second blood draw, there will be an insuline tolerance test in all patients. MRI will only be done if the last taken image is more than two years old or if the MRI was not taken with main focus on the pituitary gland.

ELIGIBILITY:
Inclusion Criteria:

* Patients that were diagnosed with an (partial) empty sella detected by MRI or CT of the brain have been included in this study. Whenever the MRI or CT scan was performed more than two years ago, a new MRI scan was required.

Exclusion Criteria:

* Children (patients less than 18 years) and patients with earlier diagnosed carcinomas of the brain as well as patients with secondary empty sella (antecedents of radiation, pharmacological treatment of pituitary adenomas, traumatic head injury and surgery of the pituitary gland as well as the central nervous system) were not included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-10-14 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients that have hormone deficiency | Within two years after empty sella has been found on MRI or CT
  The proportion of patients that have hormone deficiency when the condition "empty sella" is found on MRI or CT

CONTACTS AND LOCATIONS:
Locations (1):
- Universitair Ziekenhuis Brussel, Brussels, Jette, Belgium